CLINICAL TRIAL: NCT03531762
Title: Phase I, Open-label, Three-Period Crossover Study to Investigate the Effect of a Proton Pump Inhibitor (Omeprazole) on the PK of Tepotinib in Healthy Subjects
Brief Title: Effect of a Proton Pump Inhibitor on the PK of Tepotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200095_0039; 2017-002832-18 (EudraCT Number)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Proton Pump Inhibitor; Omeprazole; Tepotinib; Non-small cell lung cancer (NSCLC); Pharmacokinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tepotinib; Omeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1: Treatment A-B-C (Experimental): Participants received single oral dose of 500 milligrams (mg) of Tepotinib alone in fed state on Day 1 of Treatment period 1 (Treatment A) followed by single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 2 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 2 (Treatment B) followed by single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 3 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 3 (Treatment C). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole
- Sequence 2: Treatment A-C-B (Experimental): Participants received single oral dose of 500 mg of Tepotinib alone in fed state on Day 1 of Treatment period 1 (Treatment A) followed by single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 2 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 2 (Treatment C) followed by single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 3 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 3 (Treatment B). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole
- Sequence 3: Treatment B-A-C (Experimental): Participants received single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 1 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 1 (Treatment B) followed by single oral dose of 500 mg of Tepotinib alone in fed state on Day 1 of Treatment period 2 (Treatment A) followed by single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 3 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 3 (Treatment C). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole
- Sequence 4: Treatment B-C-A (Experimental): Participants received single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 1 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 1 (Treatment B) followed by single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 2 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 2 (Treatment C) followed by single oral dose of 500 mg of Tepotinib alone in fed state on Day 1 of Treatment period 3 (Treatment A). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole
- Sequence 5: Treatment C-A-B (Experimental): Participants received single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 1 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 1 (Treatment C) followed by single oral dose of 500 mg of Tepotinib alone in fed state on Day 1 of Treatment period 2 (Treatment A) followed by single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 3 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 3 (Treatment B). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole
- Sequence 6: Treatment C-B-A (Experimental): Participants received single oral dose of 500 mg Tepotinib in fed state on Day 5 of Treatment period 1 with 40 mg omeprazole once daily on Day 1 to 5 of Treatment period 1 (Treatment C) followed by single oral dose of 500 mg Tepotinib in fasted state on Day 5 of Treatment period 2 with 40 mg of omeprazole once daily on Day 1 to 5 of Treatment period 2 (Treatment B) followed by single oral dose of 500 mg of Tepotinib alone in fed state on Day 1 of Treatment period 3 (Treatment A). A washout period of at least 14 days was maintained between the Tepotinib single dose administrations.
  Interventions: Drug: Tepotinib; Drug: Omeprazole

INTERVENTIONS:
Drug: Tepotinib — Participants received single oral dose of 500 mg Tepotinib in Treatment A, B and C.
Drug: Omeprazole — Participants received omeprazole alone on Day 1 to 4 and co-administration of omeprazole with Tepotinib on Day 5 in Treatment B and C.

SUMMARY:
This study was investigated in healthy participants (i) the effect of omeprazole (proton pump inhibitor) co-administration on the single dose pharmacokinetics (PK) of tepotinib under fed conditions, and (ii) the effect of food on the single dose PK of tepotinib after co-administration of omeprazole and tepotinib. Furthermore, the study assessed the safety and tolerability of tepotinib alone and upon co-administration of omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-child bearing potential
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* Body weight between 50 to 100 kilogram (kg)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical study within 60 days prior to first drug administration
* Whole blood donation or loss of greater than (>) 450 milliliter (mL) within 60 days prior to first drug administration
* Any surgical or medical condition, or any other significant disease that could interfere with the study objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0039
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 28 participants were screened for the study. Out of which 12 participants were randomized into the study.
Period: Treatment Period 1 (8-12 Days)
Arm/Group | Sequence 1: Treatment A-B-C | Sequence 2: Treatment A-C-B | Sequence 3: Treatment B-A-C | Sequence 4: Treatment B-C-A | Sequence 5: Treatment C-A-B | Sequence 6: Treatment C-B-A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (8-12 Days)
Arm/Group | Sequence 1: Treatment A-B-C | Sequence 2: Treatment A-C-B | Sequence 3: Treatment B-A-C | Sequence 4: Treatment B-C-A | Sequence 5: Treatment C-A-B | Sequence 6: Treatment C-B-A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (8-12 Days)
Arm/Group | Sequence 1: Treatment A-B-C | Sequence 2: Treatment A-C-B | Sequence 3: Treatment B-A-C | Sequence 4: Treatment B-C-A | Sequence 5: Treatment C-A-B | Sequence 6: Treatment C-B-A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants who received single oral dose of 500 mg of Tepotinib alone in fed state (Treatment A) or in fasted state with 40 mg omeprazole (Treatment B) or in fed state with 40 mg omeprazole (Treatment C) in either Treatment period 1, Treatment Period 2 or Treatment period 3.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Tepotinib in Treatment A and Treatment C
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hour post-dose on Day 1 (for Treatment A) and on Day 5 (for Treatment C)
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least 1 dose of IMP, had no clinically important protocol deviations or important events affecting PK, and provided at least 1 measurable post dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Groups:
- Treatment A: Participants received single oral dose of Tepotinib 500 mg alone in fed state on Day 1 in either Treatment period 1 or 2 or 3.
- Treatment C: Participants received single oral dose of 500 mg of Tepotinib in fed state on Day 5 with 40 mg omeprazole once daily on Day 1 to 5 of either Treatment period 1 or 2 or 3.
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 12 | 12
Hour*nanogram per milliliter (h*ng/mL) | 21722 (18.3) | 23649 (19.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other; Ratio of Geometric Least Square Mean = 108.87, 90% CI 2-sided [101.20 to 117.13]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib in Treatment A and Treatment C
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/Lambda z, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: The PK Analysis Set included all participants who received at least 1 dose of IMP, had no clinically important protocol deviations or important events affecting PK, and provided at least 1 measurable post dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 12 | 12
h*ng/mL | 23081 (19.8) | 25343 (21.3)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other; Ratio of Geometric Least Square Mean = 109.80, 90% CI 2-sided [101.69 to 118.55]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib in Treatment A and Treatment C
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 12 | 12
Nanogram per milliliter (ng/mL) | 428 (12.2) | 445 (21.1)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other; Ratio of Geometric Least Square Mean = 104.10, 90% CI 2-sided [92.93 to 116.61]

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Tepotinib in Treatment B
Description: as for outcome 1
Time Frame: Pre-dose, 15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hour post-dose on Day 5 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Treatment B: Participants received single oral dose of 500 mg of Tepotinib in fasted state on Day 5 with 40 mg of omeprazole once daily on Day 1 to 5 of either Treatment period 1 or 2 or 3.
Arm/Group | Treatment B
Number analyzed (Participants) | 12
h*ng/mL | 16220 (24.4)

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib in Treatment B
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 12
h*ng/mL | 17412 (27.2)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib in Treatment B
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 4
Population: PK Analysis Set included all participants who received at least 1 dose of IMP, had no clinically important protocol deviations or important events affecting PK, and provided at least 1 measurable post dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment B
Number analyzed (Participants) | 12
ng/mL | 227 (25.7)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Tepotinib in Treatments A, B and C
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hour post-dose on Day 1 (for Treatment A) and on Day 5 (for Treatment B and C)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
Hours | 8.0 [6.0 to 12.0] | 12.0 [4.0 to 48.0] | 8.0 [6.0 to 12.0]

8. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Tepotinib in Treatments A, B and C
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
hour | 32.9 [23.2 to 40.5] | 30.7 [22.4 to 50.2] | 31.7 [25.8 to 48.0]

9. Secondary Outcome: Time Prior to the First Measurable (Non-zero) Concentration (Tlag) of Tepotinib in Treatments A, B and C
Description: Time prior to the first measurable (non-zero) concentration; calculated as last time point at which the concentration is less than (<) Lower Limit of Quantification (LLOQ) before the occurrence of the first quantifiable concentration.
Time Frame: as for outcome 7
Population: None of the participants were analyzed and no data was collected for this outcome as Tlag was included in the Statistical Analysis Plan and protocol in error and this parameter was not relevant for decision making. Hence, no analysis was conducted for this outcome.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Tepotinib in Treatments A, B and C
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
Liter per hour (L/h) | 19.5 (19.8) | 25.8 (27.2) | 17.8 (21.3)

11. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) of Tepotinib in Treatments A, B and C
Description: Vz/f is defined as the distribution of a study drug between plasma and the rest of the body after oral dosing.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
Liters | 912 (18.4) | 1181 (21.7) | 860 (21.9)

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether/not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 7 for Treatment A and up to Day 11 for Treatment B and C
Population: The Safety Analysis Set included all participants who received at least 1 dose of planned IMP and had 1 subsequent safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
Participants | 1 | 3 | 1

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters, 12-lead Electrocardiogram (ECG) Findings and Vital Signs
Description: The laboratory measurements included hematology, biochemistry, virology, drugs of abuse, hormones, and urinalysis. ECG recordings included PR, QRS, RR, QT and corrected QT intervals (QTcF). Vital sign assessment included blood pressure, pulse rate, body temperature. Number of participants with clinically significant abnormalities in laboratory parameters, 12-lead ECG findings, vital signs were reported. Clinically significance was decided by investigator.
Time Frame: Baseline up to Day 4 for Treatment A and up to Day 8 for Treatment B and C
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Laboratory Parameters | 0 | 0 | 0
  12-lead Electrocardiogram (ECG) Findings | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 7 for Treatment A and up to Day 11 for Treatment B and C
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=12) | Treatment B (N=12) | Treatment C (N=12)
Conjunctival cyst (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03531762/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03531762/SAP_001.pdf